CLINICAL TRIAL: NCT00907595
Title: Treating Sleep Wake Cycle Disturbances in Basal Ganglia Neurodegenerative Disorder Subjects With Ramelteon- A Double Blind, Placebo Controlled Trial
Brief Title: Treating Sleep/Wake Cycle Disturbances in Basal Ganglia Disorders With Ramelteon
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to recruit subjects for study.Collaborator stopped funding for study as of 3/31/2010
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Kaloyan Tanev, MD, Neuropsychiatrist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-043R
Record Dates: First submitted 2009-05-20; First posted 2009-05-22 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: Huntington's Disease; Parkinson's Disease; Dementia With Lewy Bodies; Sleep Disorders; Circadian Dysregulation
Keywords: Huntington's chorea; Huntington's Disease; Parkinson's Disease; Parkinsonism; Dementia; Dementia with Lewy Bodies; Actigraphy; Circadian dysregulation; Sleep Disorders; Circadian rhythm
MeSH Terms: conditions — Huntington Disease; Parkinson Disease; Lewy Body Disease; Sleep Wake Disorders; Chronobiology Disorders; Parkinsonian Disorders; Dementia | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ramelteon (Active Comparator): Subjects randomized to Ramelteon
  Interventions: Drug: Ramelteon
- Placebo (Placebo Comparator): Subjects randomized to placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ramelteon — After 2 weeks of baseline sleep study, subjects will be randomized to take either Ramelteon or Placebo for 4 weeks.
  Arms: Ramelteon
Drug: Placebo — After 2 weeks of baseline sleep study, subjects will be randomized to take either Ramelteon or Placebo for 4 weeks.
  Arms: Placebo

SUMMARY:
The proposed study is a double-blind, placebo controlled pilot study of HD, PD, and DLB subjects with sleep disturbances. This study is designed to determine the effects of 4 weeks Ramelteon treatment on the sleep patterns of people with basal ganglia disorders such as HD, PD and DLB. The study also aims to look at the sleep patterns of caregivers of people with HD, PD and DLB.

DETAILED DESCRIPTION:
Huntington's disease (HD) is a progressively degenerative brain disorder, which results in a loss of mental and physical abilities. It is genetically determined and people carrying the HD gene invariably develop the clinical disorder at some point in their lives. HD symptoms consist of neuropsychiatric changes and motor movements. Once present, the symptoms are progressive in nature and eventually fatal. Currently there is no cure for HD.

Like HD, Parkinson's Disease (PD) and Dementia with Lewy Bodies (DLB) are also neurodegenerative disorders affecting the basal ganglia. PD and DLB are synucleinopathies - i.e., they are associated with dysfunction of the protein alpha-synuclein. Unlike HD, PD and DLB are not inherited in an autosomal dominant manner.

Sleep/wake cycles in HD, PD and DLB. HD patients, especially those in moderate to severe stages of the disease, frequently complain of difficulty falling and staying asleep. Little is known about the phenomenology and pathophysiology of sleep disturbances in HD. The few studies that have addressed this issue of sleep in HD have found disturbances in sleep architecture and sleep/wake cycles. Overall, the literature on sleep and other circadian disturbances in HD is very limited. If sleep/wake cycle disturbances in HD have pathophysiological mechanisms similar to other neurodegenerative disorders, then Ramelteon, a hypnotic agent and melatonin receptor agonist, may be beneficial in sleep/wake cycle disturbances in HD.

Sleep disruptions and circadian sleep disruptions are integral to the clinical presentation of both PD and DLB. As is true in HD, sleep disturbances in PD and DLB cause severe disruption to the patients and their caregivers' lives. In PD, sleep dysfunction occurs in approximately two thirds of patients. Sleep problems range from difficulty with sleep initiation, sleep fragmentation, disturbance of circadian rhythm, REM sleep behavior disorder (RBD), to excessive daytime sleepiness. Frequent nighttime awakening and sleep disruption are the most common sleep problems in PD. In DLB, REM sleep behavior disorder (RBD) occurs years to decades before the onset of dementia. Importantly, melatonin is one of the main treatments used for RBD. Therefore, a melatonin agonist such as Ramelteon is a natural choice for the treatment of circadian sleep disturbances in PD and DLB.

Activity monitors (actigraphs) have been used as an alternative to polysomnography (PSG). Actigraphs are small electronic motion sensors that detect movements in three axes and provide information about the subjects' activity levels over periods of days to weeks. Using validated algorithms to infer wakefulness and sleep, investigators can draw conclusions about the individuals' sleep/wake cycle patterns from their activity patterns.

ELIGIBILITY:
We will recruit 24 Huntington's disease, Parkinson's Disease, or Dementia with Lewy Bodies subjects. Assuming a dropout rate of 20%, we expect that 20 of the 24 subjects who initially enroll will complete the study.

Inclusion criteria will be the following:

* Subjects with HD will be between the ages of 20 and 65 years old;
* Subjects with PD or DLB will be between the ages of 40 and 90;
* Subjects will have subjective complaints of sleeping problems or their caregivers will complain of the subjects not sleeping well
* Subjects with all severity of HD, PD, and DLB symptoms will be accepted as long as they complain of sleep problems
* A diagnosis of HD, PD, or DLB. For HD patients, a positive HD gene status for everyone except the caregivers will have been obtained for clinical reasons and will be known at the time of enrollment into the study. PD patients will have a clinical diagnosis of PD. DLB patients will have a diagnosis of possible or probably DLB based on consensus criteria (outlined in McKeith et al., 2005).
* Subjects will be willing and able to participate in the informed consent process.

Exclusion criteria will be the following:

* Subjects who are unable to participate in the informed consent process
* Subjects with previously documented primary sleep disorders (unrelated to HD, PD, or DLB), including Obstructive Sleep Apnea Syndrome, Periodic Limb Movement Disorder of Sleep, or Narcolepsy.
* Subjects taking fluvoxamine, rifampin, ketoconazole , and fluconazole within 30 days of baseline
* Subjects with hepatic impairment
* Subjects who perform shift work or have any other circadian rhythm abnormality or disruption
* Subjects who are diagnosed with a Major Depressive Episode, current at the time of enrollment (subject may have a history of a Major Depressive Episode as long as it is in partial or full remission at the time of enrollment)
* Subjects who are diagnosed with a manic or hypomanic episode, current at the time of enrollment (subject may have a history of a manic or hypomanic episode as long as it is in full remission at the time of enrollment)
* Subjects who at the time of enrollment receive hypnotic agents or have been on hypnotic agents during the two weeks prior to enrollment
* Subjects who are pregnant at the time of enrollment or intend to become pregnant during the period of study participation
* Subjects who in the opinion of the research personnel would not be able to participate in the research protocol because of agitation, lack of transportation, or other reasons.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-05; Primary Completion 2010-03 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Sleep efficiency and other actigraphy derived sleep parameters | 2 weeks pre intervention; 4 weeks of the intervention; 2 weeks after intervention

SECONDARY OUTCOMES:
UHDRS, UPDRS, cognitive measures, mood symptoms, aggression measures, functional ability. | 2 weeks pre intervention; 4 weeks of the intervention; 2 weeks after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Kaloyan S Tanev, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Hurelbrink CB, Lewis SJ, Barker RA. The use of the Actiwatch-Neurologica system to objectively assess the involuntary movements and sleep-wake activity in patients with mild-moderate Huntington's disease. J Neurol. 2005 Jun;252(6):642-7. doi: 10.1007/s00415-005-0709-z. Epub 2005 Mar 7. PMID 15742112
- [Background] Morton AJ, Wood NI, Hastings MH, Hurelbrink C, Barker RA, Maywood ES. Disintegration of the sleep-wake cycle and circadian timing in Huntington's disease. J Neurosci. 2005 Jan 5;25(1):157-63. doi: 10.1523/JNEUROSCI.3842-04.2005. PMID 15634777
- [Background] Ancoli-Israel S, Clopton P, Klauber MR, Fell R, Mason W. Use of wrist activity for monitoring sleep/wake in demented nursing-home patients. Sleep. 1997 Jan;20(1):24-7. doi: 10.1093/sleep/20.1.24. PMID 9130330